CLINICAL TRIAL: NCT04957381
Title: The Effect of Cardiopulmonary and Muscular Fitness on Healthy Aging Among Community-Dwelling Older Adults
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Mei-Wun Tsai, Associate professor, National Yang Ming Chiao Tung University
Other Study IDs: YM109154E
Record Dates: First submitted 2021-04-26; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Healthy Aging
Keywords: Healthy aging; Cardiorespiratory fitness; Muscular fitness; Health promotion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- low to moderate CRF with low MF: According to the senior fitness test norms in Taiwan, participants with low to moderate cardiorespiratory fitness (CRF) and low muscular fitness (MF).
  Interventions: Behavioral: Group exercises
- low to moderate CRF with moderate MF: According to the senior fitness test norms in Taiwan, participants with low to moderate cardiorespiratory fitness (CRF) and moderate muscular fitness (MF).
  Interventions: Behavioral: Group exercises
- low to moderate CRF with high MF: According to the senior fitness test norms in Taiwan, participants with low to moderate cardiorespiratory fitness (CRF) and high muscular fitness (MF).
  Interventions: Behavioral: Group exercises
- high CRF with low to moderate MF: According to the senior fitness test norms in Taiwan, participants with high cardiorespiratory fitness (CRF) and low to moderate muscular fitness (MF).
  Interventions: Behavioral: Group exercises
- high CRF and high MF: According to the senior fitness test norms in Taiwan, participants with high cardiorespiratory fitness (CRF) and high muscular fitness (MF).
  Interventions: Behavioral: Group exercises

INTERVENTIONS:
Behavioral: Group exercises — Group exercises including aerobic, resistance and stretching exercise. Once a week for 8-12 weeks.

SUMMARY:
To compare the different cardiopulmonary and muscular fitness of community-dwelling older adults on healthy aging, and to identify the optimal cutoff points of their cardiopulmonary fitness and muscular fitness on targeting healthy aging.

DETAILED DESCRIPTION:
At the end of the 20th century, the WHO began to promote the issue of healthy aging. From then on, the Taiwan government gradually attached importance to long-term care and devoted to developing community-based health promotion programs for the elderly. Currently, the programs commonly plan to proceed through the group exercise intervention, increasing physical activity to improve their physical fitness and also to prevent their functional disability. This study aims to compare the different cardiorespiratory fitness and muscular fitness of community-dwelling older adults on healthy aging, and figure out to what extent of cardiorespiratory fitness level and muscular fitness level may achieve healthy aging. The present healthy status of participants will be investigated by interviewing if having any disability or frail. Based on multidimensional model, the definition and measurement of healthy aging status include physiological, psychological and social function aspect. In this study, the health aging status is defined as non-frailty, independence in basic and instrumental activities of daily living, normal cognitive function, absent of depression status, good social relations and good environmental support.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 55 years old
* Had contact information from project
* Had attended both pre-test or post-test during program
* Volunteer to participant

Exclusion Criteria:

* Incomplete physical fitness data
* Participant with frailty after screening during the class
* Not available to respond
* Not accept the informed consent

Ages: 55 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older adults
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-11-11 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Physiological health: non-frailty | once follow up at 2-4 years after community-based health promotion programs
  SOF index (study of osteoporotic fracture index). Minimum value is 0 and maximum value is 3. Non-frailty is defined as the score less than 2 points.
Physiological health: independence in basic activities of daily living | once follow up at 2-4 years after community-based health promotion programs
  Katz ADL index (Katz index of independence in activities of daily living). Minimum value is 0 and maximum value is 6. Independence in basic ADL is defined as that score 0 point.
Physiological health: independence in instrumental activities of daily living | once follow up at 2-4 years after community-based health promotion programs
  Lawton IADL scale (Lawton scale of instrumental activities of daily living). Minimum value is 0 and maximum value is 8. Independence in IADL is defined as that score 0 point.
Mental health: normal cognitive function | once follow up at 2-4 years after community-based health promotion programs
  MoCA (Montreal cognitive assessment). Minimum value is 0 and maximum value is 30. Normal cognitive function is defined as score above 24.
Mental health: absent of depression status | once follow up at 2-4 years after community-based health promotion programs
  GDS-15 (short form geriatric depression scale). Minimum value is 0 and maximum value is 15. Absent of depression status is defined as score less than 5.
Social function: good social relations | once follow up at 2-4 years after community-based health promotion programs
  WHOQOL-BREF (WHO Quality of Life-BREF questionnaire). Minimum value is 4 and maximum value is 20. Good social relations is defined as score above 15.
Social function: good environmental support | once follow up at 2-4 years after community-based health promotion programs
  WHOQOL-BREF (WHO Quality of Life-BREF questionnaire). Minimum value is 4 and maximum value is 20. Good environment support is defined as score above 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Tsai, Mei-Wun, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided